CLINICAL TRIAL: NCT02419911
Title: Prospective, Randomized Comparison of the Use of FloShield Air System Versus Clearify Visualization System (D-HELP) During Laparoscopic Surgery to Evaluate the Operative Interruption for Lens Cleaning
Brief Title: Comparison FloShield Air System Versus Clearify Visualization System (D-HELP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Minimally Invasive Devices, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: FSA-0001
Record Dates: First submitted 2015-04-01; First posted 2015-04-17 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-05

CONDITIONS: Laparoscopic Surgery
Keywords: gastrointestinal; gynecologic; urologic; bariatric; laparoscopic surgery
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FloShield (Other): FloShield Air Laparoscopic Cleaning and Defogging System used during laparoscopic surgery
  Interventions: Procedure: Laparoscopic surgery; Device: FloShield Defogging and Cleaning System
- Clearify (Other): Clearify Visualization System used during laparoscopic surgery
  Interventions: Procedure: Laparoscopic surgery; Device: Clearify Defogging and Cleaning System

INTERVENTIONS:
Procedure: Laparoscopic surgery — gastrointestinal, gynecologic, urologic or bariatric laparoscopic surgery;
Device: FloShield Defogging and Cleaning System — Sterile, single-use in vivo device to clean and defog the laparoscope camera lens
  Other Names: FloShield System
  Arms: FloShield
Device: Clearify Defogging and Cleaning System — Single-use, ex vivo device to clean and defog the laparoscope camera lens
  Arms: Clearify

SUMMARY:
This is a post market, prospective, comparison study of the use of the FloShield Air System versus Clearify™ Visualization System (D-HELP) during laparoscopic surgery.

DETAILED DESCRIPTION:
This is a post market, prospective, comparison study of the use of the FloShield Air System versus Clearify™ Visualization System (D-HELP) during laparoscopic surgery. The study will be randomized across two groups, one group will evaluate laparoscopic lens cleaning with D-HELP during laparoscopic surgery and the second group will evaluate laparoscopic lens cleaning using the FloShield Air System during laparoscopic surgery. Each surgery will be captured on video. Study parameters will be evaluated through review of each video by an independent evaluator.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male;
* 18 years of age or older;
* Patient scheduled for gastrointestinal, gynecologic, urologic or bariatric laparoscopic surgery under the care of the study investigator;
* Suitable candidate for surgery

Exclusion Criteria:

* Unfit for surgery: concomitant disorders incompatible with the study or surgery (at the discretion of the investigator);
* Use of Surgiquest AirSeal®;
* Use of humidified insufflation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
number of Laparoscope removals during surgery | 0.5hr - 6hr
  The performance evaluations of the FloShield Air System will be based the difference between the cohorts on the number of scope removals per surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Poll, MD, Study Director — President and CEO
Locations (3):
- United States (3):
  - South Miami Hospital, South Miami, Florida
  - Centennial Hills Medical Center, Las Vegas, Nevada
  - University of Cincinnati, Cincinnati, Ohio